CLINICAL TRIAL: NCT06369246
Title: PRORAD-5 PROstate RADiation in 5 Fractions: Phase Ib Five Fraction Radiotherapy for Patients With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0893; NCI-2024-03308 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental): Participants will then be scheduled to receive radiation therapy. Radiation will be given over 5 sessions, 2-3 times per week, for 2 weeks. Each radiation therapy session will take 15-30 minutes to complete.
  Within 1 day after completing radiation therapy, blood (about 2 tablespoons) will be drawn for routine tests.
  Interventions: Device: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Device: Stereotactic Body Radiation Therapy — Undergo Radiation Therapy

SUMMARY:
To look at the safety and effectiveness of stereotactic body radiation therapy (SBRT) in treating advanced or high-risk prostate cancer.

DETAILED DESCRIPTION:
Primary Objectives:

Primary Objective #1: To determine the proportion of patients experiencing late grade ≥ 3 GI toxicity after five fraction pelvic nodal RT as reported by the treating physician at 3 months post-treatment.

Primary Objective #2: To estimate the change in health-related quality of life (HRQOL) following the proposed treatment regimen compared to pre-treatment assessment 6 months after completing RT. Patient-reported urinary, bowel, and sexual function and general QoL will be collected using validated EPIC-26, EQ-5D, PROMIS-Fatigue questionnaires prior to RT, at the end of RT 3, and 6, 12, 24 months after completion of RT.

Secondary Objectives:

Secondary Objective #1: To estimate the metastasis free survival (MFS) at 24 months after study enrollment. All time-to-event analyses will be analyzed indexed to date of study enrollment.

Secondary Objective #2: To estimate the rate of acute and late GI and GU toxicity of the treatment regimen

Secondary Objective #3: To assess adherence to protocol treatment parameters. RT plans will be evaluated for contouring consistency, target coverage and tissue constraint adherence with the use of artificial intelligence (AI) auto-segmentation/contours and scorecards to facilitate this process and improve plan quality and clinical efficiency.

Secondary Objective #4: To explore the impact of five fraction pelvic nodal RT on lymphopenia.

White blood cell counts will be obtained before and after treatment and compared to historical data on lymphopenia with conventionally fractionated pelvic RT.

Secondary Objective #5: To estimate HRQOL following the proposed treatment regimen compared to pre-treatment assessment at the end of RT 3 months, 12, and 24 months after completing RT and assess the HRQOL change over time.

Exploratory Objective #1: To investigate the effect of pelvic nodal RT on gut microbiome with gut microbiome sample collection pre- and upon RT completion.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma of prostate within one year of study entry. Evaluation can happen outside of MD Anderson as long as histological confirmation takes place at MD Anderson.

   1. cT1c-T3a by digital exam or imaging (AJCC 8th Ed.). No cT3b-4 by digital exam or imaging (AJCC 8th Ed.)
   2. Gleason Grade Group 2-5 (Gleason 7, 8, 9, 10).
   3. If Gleason Grade 2, must meet definition of unfavorable intermediate risk (at least one of the following: cT2b, PSA >10 ng/mL prior to starting androgen deprivation therapy (ADT).

   If a participant is taking 5-alpha reductase inhibitors the measured PSA may be doubled).
2. Node negative by conventional imaging.
3. Be ≥ 18 years of age on the day of signing informed consent.
4. Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation (both LHRH agonist and oral anti-androgen) is ≤ 185 days prior to registration; Please note: baseline PSA must be obtained prior to the start of any ADT.
5. ECOG performance status 0-2.

Exclusion Criteria:

1. Diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe RT.
2. Prior prostatectomy, cryosurgery, or HIFU for adenocarcinoma of the prostate
3. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields
4. Distant metastatic disease on conventional imaging, which by the discretion of the treating physician cannot be treated definitively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Comron Hassanzadeh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org